CLINICAL TRIAL: NCT01123486
Title: A Hydromorphone High Resolution Pharmacokinetic-Pharmacodynamic Fingerprint as the Basis for Identifying Sex Differences in Opioid Pharmacokinetics and Pharmacodynamics
Brief Title: Hydromorphone Pharmacokinetic-Pharmacodynamic Fingerprint
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI relocated to new university
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dhanesh Gupta, Associate Professor of Anesthesiology & Neurological Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00013543
Record Dates: First submitted 2010-05-10; First posted 2010-05-14 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Pain; Ventilatory Depression
Keywords: Intravenous opioids; Patient Controlled Analgesia; volunteer pharmacokinetic-pharmacodynamic study
MeSH Terms: conditions — Pain; Respiratory Insufficiency | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hydromorphone (Experimental): open label single arm pharmacokinetic-pharmacodynamic study
  Interventions: Drug: hydromorphone

INTERVENTIONS:
Drug: hydromorphone — hydromorphone 0.02 mg/kg
  Other Names: Dilaudid

SUMMARY:
The primary objective of the proposed work is development of a high resolution pharmacokinetic-pharmacodynamic (PK-PD) model of hydromorphone for experimental pain stimuli, ventilatory depression, and surrogate biomarkers of opioid effect that will allow the fingerprinting of hydromorphone. This fingerprint will serve as the basis for the development of dosing strategies that efficiently maximize analgesia while minimizing ventilatory depression and sedation. For example, this high-resolution fingerprint will allow precise estimation of an initial hydromorphone target effect site concentration (Ce) from those of effectively administered synthetic opioids with previously determined high-resolution fingerprints (i.e., remifentanil or fentanyl), thereby minimizing underdosing of hydromorphone for analgesia and minimizing side effects.

DETAILED DESCRIPTION:
After 6 h of fasting, each volunteer will have a 20G arterial-line placed in the radial artery for early blood sampling and an 18 G peripheral intravenous catheter placed in the contralateral forearm for drug administration and later blood sampling. Continuously monitored vital signs will include ECG, invasive blood pressure, hemoglobin, O2 saturation, end-tidal CO2, and respiratory rate (from the capnogram) recorded.

After baseline PD data acquisition, a bolus of 0.2 mg/kg hydromorphone will be administered over 10 sec via the free-flowing peripheral IV (t=0) and 3 mL arterial blood samples will be obtained at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, and 2 min using a stop-cock and manifold system. Subsequent blood samples will be acquired at 3, 4, 5, 7.5, 10, 15, 20, 25, 30, and 45 min and 1, 1.25, 1.5, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 20, and 24 h. Although EEG will be acquired continuously, the remaining pharmacologic data will be recorded at discrete times s in the initial 5 min: pupillometry at 1, 2, and 5 min; ventilation at 2 min; temperature analgesia at 3 and 5 min, and sedation level at 4 min. This will allow the ventilation and pupillometry to be acquired in a resting state, thereby limiting distortion of these responses by stimulation. Subsequently, all data will be acquired at all PK time points in the following sequence - ventilation and EEG (simultaneously), pupillometry, modified OAA/S score, and temperature analgesia. After 2 h, once a pharmacologic parameter has returned to baseline for 2 sequential measurements, recording of that parameter will be stopped. During the study, if the volunteer is unable to use the device trigger, due to opioid-induced sedation, the tolerance level for increased temperature will be defined as the temperature at which the volunteer exhibits withdrawal movement of the tested limb. Once all data acquisition has been completed, the volunteer will be allowed to drink clear liquids. Subsequently, the diet will be advanced as tolerated. The volunteer will be monitored hourly (vital signs) in the Clinical Research Unit until all of the blood samples have been acquired.

ELIGIBILITY:
Inclusion Criteria:

* within 20% of their ideal body weight
* 21-30 years old
* ASA I (no systemic disease)
* No history of PONV (except wisdom teeth extraction)
* No long term medication use
* No history of coagulation defect (i.e easy bruising, gum bleeding with teeth brushing, frequent nose bleeds, past documented coagulopathy, etc.)

Exclusion Criteria:

* Inability to place an arterial line
* A failed urine drug test on admission to the CRU
* A positive pregnancy test on admission to the CRU
* A hemoglobin level < 12.5 g/dL on admission to the CRU

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Opioid induced analgesia | 24 hours
  A combined PK-PD model for hydromorphone induced analgesia (heat pain tolerance) will be developed

SECONDARY OUTCOMES:
Opioid induced ventilatory depression | 24 hours
  A combined PK-PD model for hydromorphone induced ventilatory depression will be created
Opioid induced miosis | 24 hours
  A combined PK-PD model for hydromorphone induced miosis will be developed
Opioid induced EEG changes | 24 hours
  A combined PK-PD model for hydromorphone induced EEG effects will be developed

CONTACTS AND LOCATIONS:
Overall Officials: Dhanesh K. Gupta, M.D., Principal Investigator — Departments of Anesthesiology & Neurological Surgery, Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Upton RN, Semple TJ, Macintyre PE. Pharmacokinetic optimisation of opioid treatment in acute pain therapy. Clin Pharmacokinet. 1997 Sep;33(3):225-44. doi: 10.2165/00003088-199733030-00005. PMID 9314613
- [Background] Stanski DR, Hug CC Jr. Alfentanil--a kinetically predictable narcotic analgesic. Anesthesiology. 1982 Dec;57(6):435-8. doi: 10.1097/00000542-198212000-00001. No abstract available. PMID 6128947
- [Background] Scott JC, Ponganis KV, Stanski DR. EEG quantitation of narcotic effect: the comparative pharmacodynamics of fentanyl and alfentanil. Anesthesiology. 1985 Mar;62(3):234-41. doi: 10.1097/00000542-198503000-00005. PMID 3919613
- [Background] Maitre PO, Vozeh S, Heykants J, Thomson DA, Stanski DR. Population pharmacokinetics of alfentanil: the average dose-plasma concentration relationship and interindividual variability in patients. Anesthesiology. 1987 Jan;66(1):3-12. PMID 3099604
- [Background] Scott JC, Stanski DR. Decreased fentanyl and alfentanil dose requirements with age. A simultaneous pharmacokinetic and pharmacodynamic evaluation. J Pharmacol Exp Ther. 1987 Jan;240(1):159-66. PMID 3100765
- [Background] Scott JC, Cooke JE, Stanski DR. Electroencephalographic quantitation of opioid effect: comparative pharmacodynamics of fentanyl and sufentanil. Anesthesiology. 1991 Jan;74(1):34-42. doi: 10.1097/00000542-199101000-00007. PMID 1670913
- [Background] Bjorkman S, Wada DR, Stanski DR, Ebling WF. Comparative physiological pharmacokinetics of fentanyl and alfentanil in rats and humans based on parametric single-tissue models. J Pharmacokinet Biopharm. 1994 Oct;22(5):381-410. doi: 10.1007/BF02353862. PMID 7791038
- [Background] Egan TD, Minto CF, Hermann DJ, Barr J, Muir KT, Shafer SL. Remifentanil versus alfentanil: comparative pharmacokinetics and pharmacodynamics in healthy adult male volunteers. Anesthesiology. 1996 Apr;84(4):821-33. doi: 10.1097/00000542-199604000-00009. PMID 8638836
- [Background] Minto CF, Schnider TW, Egan TD, Youngs E, Lemmens HJ, Gambus PL, Billard V, Hoke JF, Moore KH, Hermann DJ, Muir KT, Mandema JW, Shafer SL. Influence of age and gender on the pharmacokinetics and pharmacodynamics of remifentanil. I. Model development. Anesthesiology. 1997 Jan;86(1):10-23. doi: 10.1097/00000542-199701000-00004. PMID 9009935
- [Background] Minto CF, Schnider TW, Shafer SL. Pharmacokinetics and pharmacodynamics of remifentanil. II. Model application. Anesthesiology. 1997 Jan;86(1):24-33. doi: 10.1097/00000542-199701000-00005. PMID 9009936
- [Background] Egan TD, Lemmens HJ, Fiset P, Hermann DJ, Muir KT, Stanski DR, Shafer SL. The pharmacokinetics of the new short-acting opioid remifentanil (GI87084B) in healthy adult male volunteers. Anesthesiology. 1993 Nov;79(5):881-92. doi: 10.1097/00000542-199311000-00004. PMID 7902032
- [Background] Segre G. Kinetics of interaction between drugs and biological systems. Farmaco Sci. 1968 Oct;23(10):907-18. No abstract available. PMID 5712792
- [Background] Sheiner LB, Stanski DR, Vozeh S, Miller RD, Ham J. Simultaneous modeling of pharmacokinetics and pharmacodynamics: application to d-tubocurarine. Clin Pharmacol Ther. 1979 Mar;25(3):358-71. doi: 10.1002/cpt1979253358. PMID 761446
- [Background] Ebling WF, Lee EN, Stanski DR. Understanding pharmacokinetics and pharmacodynamics through computer stimulation: I. The comparative clinical profiles of fentanyl and alfentanil. Anesthesiology. 1990 Apr;72(4):650-8. doi: 10.1097/00000542-199004000-00013. PMID 2321782
- [Background] Gregg KM, Varvel JR, Shafer SL. Application of semilinear canonical correlation to the measurement of opioid drug effect. J Pharmacokinet Biopharm. 1992 Dec;20(6):611-35. doi: 10.1007/BF01064422. PMID 1302765
- [Background] Lemmens HJ, Dyck JB, Shafer SL, Stanski DR. Pharmacokinetic-pharmacodynamic modeling in drug development: application to the investigational opioid trefentanil. Clin Pharmacol Ther. 1994 Sep;56(3):261-71. doi: 10.1038/clpt.1994.136. PMID 7924121
- [Background] Lemmens HJ, Egan TD, Fiset P, Stanski DR. Pharmacokinetic/dynamic assessment in drug development: application to the investigational opioid mirfentanil. Anesth Analg. 1995 Jun;80(6):1206-11. doi: 10.1097/00000539-199506000-00024. PMID 7762853
- [Background] Kern SE, Stanski DR. Pharmacokinetics and pharmacodynamics of intravenously administered anesthetic drugs: concepts and lessons for drug development. Clin Pharmacol Ther. 2008 Jul;84(1):153-7. doi: 10.1038/clpt.2008.80. Epub 2008 May 7. PMID 18463623
- [Background] Ausems ME, Vuyk J, Hug CC Jr, Stanski DR. Comparison of a computer-assisted infusion versus intermittent bolus administration of alfentanil as a supplement to nitrous oxide for lower abdominal surgery. Anesthesiology. 1988 Jun;68(6):851-61. doi: 10.1097/00000542-198806000-00004. PMID 3132059
- [Background] Maitre PO, Ausems ME, Vozeh S, Stanski DR. Evaluating the accuracy of using population pharmacokinetic data to predict plasma concentrations of alfentanil. Anesthesiology. 1988 Jan;68(1):59-67. doi: 10.1097/00000542-198801000-00010. PMID 3122601
- [Background] Maitre PO, Stanski DR. Bayesian forecasting improves the prediction of intraoperative plasma concentrations of alfentanil. Anesthesiology. 1988 Nov;69(5):652-9. doi: 10.1097/00000542-198811000-00004. PMID 3142308
- [Background] Raemer DB, Buschman A, Varvel JR, Philip BK, Johnson MD, Stein DA, Shafer SL. The prospective use of population pharmacokinetics in a computer-driven infusion system for alfentanil. Anesthesiology. 1990 Jul;73(1):66-72. doi: 10.1097/00000542-199007000-00011. PMID 2360742
- [Background] Shafer SL, Varvel JR, Aziz N, Scott JC. Pharmacokinetics of fentanyl administered by computer-controlled infusion pump. Anesthesiology. 1990 Dec;73(6):1091-102. doi: 10.1097/00000542-199012000-00005. PMID 2248388
- [Background] Shafer SL, Varvel JR. Pharmacokinetics, pharmacodynamics, and rational opioid selection. Anesthesiology. 1991 Jan;74(1):53-63. doi: 10.1097/00000542-199101000-00010. PMID 1824743
- [Background] Shafer SL, Gregg KM. Algorithms to rapidly achieve and maintain stable drug concentrations at the site of drug effect with a computer-controlled infusion pump. J Pharmacokinet Biopharm. 1992 Apr;20(2):147-69. doi: 10.1007/BF01070999. PMID 1629794
- [Background] Fiset P, Mathers L, Engstrom R, Fitzgerald D, Brand SC, Hsu F, Shafer SL. Pharmacokinetics of computer-controlled alfentanil administration in children undergoing cardiac surgery. Anesthesiology. 1995 Nov;83(5):944-55. doi: 10.1097/00000542-199511000-00006. PMID 7486179
- [Background] Hughes MA, Glass PS, Jacobs JR. Context-sensitive half-time in multicompartment pharmacokinetic models for intravenous anesthetic drugs. Anesthesiology. 1992 Mar;76(3):334-41. doi: 10.1097/00000542-199203000-00003. PMID 1539843
- [Background] Shafer SL, Stanski DR. Improving the clinical utility of anesthetic drug pharmacokinetics. Anesthesiology. 1992 Mar;76(3):327-30. doi: 10.1097/00000542-199203000-00001. No abstract available. PMID 1539841
- [Background] Dahan A, Romberg R, Teppema L, Sarton E, Bijl H, Olofsen E. Simultaneous measurement and integrated analysis of analgesia and respiration after an intravenous morphine infusion. Anesthesiology. 2004 Nov;101(5):1201-9. doi: 10.1097/00000542-200411000-00021. PMID 15505457
- [Background] Dershwitz M, Walsh JL, Morishige RJ, Connors PM, Rubsamen RM, Shafer SL, Rosow CE. Pharmacokinetics and pharmacodynamics of inhaled versus intravenous morphine in healthy volunteers. Anesthesiology. 2000 Sep;93(3):619-28. doi: 10.1097/00000542-200009000-00009. PMID 10969293
- [Background] Coda B, Tanaka A, Jacobson RC, Donaldson G, Chapman CR. Hydromorphone analgesia after intravenous bolus administration. Pain. 1997 May;71(1):41-8. doi: 10.1016/s0304-3959(97)03336-8. PMID 9200172
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Pharmacodynamics and pharmacokinetics of methadone during the perioperative period. Anesthesiology. 1982 Dec;57(6):458-67. doi: 10.1097/00000542-198212000-00005. No abstract available. PMID 6128949
- [Background] Ausems ME, Hug CC Jr, Stanski DR, Burm AG. Plasma concentrations of alfentanil required to supplement nitrous oxide anesthesia for general surgery. Anesthesiology. 1986 Oct;65(4):362-73. doi: 10.1097/00000542-198610000-00004. PMID 3094407
- [Background] Bouillon T, Bruhn J, Radu-Radulescu L, Andresen C, Cohane C, Shafer SL. A model of the ventilatory depressant potency of remifentanil in the non-steady state. Anesthesiology. 2003 Oct;99(4):779-87. doi: 10.1097/00000542-200310000-00007. PMID 14508307
- [Background] Vuyk J, Lim T, Engbers FH, Burm AG, Vletter AA, Bovill JG. Pharmacodynamics of alfentanil as a supplement to propofol or nitrous oxide for lower abdominal surgery in female patients. Anesthesiology. 1993 Jun;78(6):1036-45; discussion 23A. doi: 10.1097/00000542-199306000-00005. PMID 8512096
- [Background] Billard V, Gambus PL, Chamoun N, Stanski DR, Shafer SL. A comparison of spectral edge, delta power, and bispectral index as EEG measures of alfentanil, propofol, and midazolam drug effect. Clin Pharmacol Ther. 1997 Jan;61(1):45-58. doi: 10.1016/S0009-9236(97)90181-8. PMID 9024173
- [Background] Phimmasone S, Kharasch ED. A pilot evaluation of alfentanil-induced miosis as a noninvasive probe for hepatic cytochrome P450 3A4 (CYP3A4) activity in humans. Clin Pharmacol Ther. 2001 Dec;70(6):505-17. doi: 10.1067/mcp.2001.119994. PMID 11753266
- [Background] Kharasch ED, Hoffer C, Walker A, Sheffels P. Disposition and miotic effects of oral alfentanil: a potential noninvasive probe for first-pass cytochrome P4503A activity. Clin Pharmacol Ther. 2003 Mar;73(3):199-208. doi: 10.1067/mcp.2003.30. PMID 12621385
- [Background] Kharasch ED, Walker A, Hoffer C, Sheffels P. Intravenous and oral alfentanil as in vivo probes for hepatic and first-pass cytochrome P450 3A activity: noninvasive assessment by use of pupillary miosis. Clin Pharmacol Ther. 2004 Nov;76(5):452-66. doi: 10.1016/j.clpt.2004.07.006. PMID 15536460
- [Background] Baririan N, Van Obbergh L, Desager JP, Verbeeck RK, Wallemacq P, Starkel P, Horsmans Y. Alfentanil-induced miosis as a surrogate measure of alfentanil pharmacokinetics in patients with mild and moderate liver cirrhosis. Clin Pharmacokinet. 2007;46(3):261-70. doi: 10.2165/00003088-200746030-00006. PMID 17328584
- [Background] Davis JJ, Swenson JD, Hall RH, Dillon JD, Johnson KB, Egan TD, Pace NL, Niu SY. Preoperative "fentanyl challenge" as a tool to estimate postoperative opioid dosing in chronic opioid-consuming patients. Anesth Analg. 2005 Aug;101(2):389-395. doi: 10.1213/01.ANE.0000156563.25878.19. PMID 16037150
- [Background] Angst MS, Chu LF, Tingle MS, Shafer SL, Clark JD, Drover DR. No evidence for the development of acute tolerance to analgesic, respiratory depressant and sedative opioid effects in humans. Pain. 2009 Mar;142(1-2):17-26. doi: 10.1016/j.pain.2008.11.001. Epub 2009 Jan 9. PMID 19135798
- [Background] Manyam SC, Gupta DK, Johnson KB, White JL, Pace NL, Westenskow DR, Egan TD. Opioid-volatile anesthetic synergy: a response surface model with remifentanil and sevoflurane as prototypes. Anesthesiology. 2006 Aug;105(2):267-78. doi: 10.1097/00000542-200608000-00009. PMID 16871060
- [Background] Manyam SC, Gupta DK, Johnson KB, White JL, Pace NL, Westenskow DR, Egan TD. When is a bispectral index of 60 too low?: Rational processed electroencephalographic targets are dependent on the sedative-opioid ratio. Anesthesiology. 2007 Mar;106(3):472-83. doi: 10.1097/00000542-200703000-00011. PMID 17325505
- [Background] Barrett PH, Bell BM, Cobelli C, Golde H, Schumitzky A, Vicini P, Foster DM. SAAM II: Simulation, Analysis, and Modeling Software for tracer and pharmacokinetic studies. Metabolism. 1998 Apr;47(4):484-92. doi: 10.1016/s0026-0495(98)90064-6. PMID 9550550
- [Background] Kuipers JA, Boer F, Olofsen E, Bovill JG, Burm AG. Recirculatory pharmacokinetics and pharmacodynamics of rocuronium in patients: the influence of cardiac output. Anesthesiology. 2001 Jan;94(1):47-55. doi: 10.1097/00000542-200101000-00012. PMID 11135721